CLINICAL TRIAL: NCT05595798
Title: Associations Between Breath Sound Frequency Pattern, Capnography and Electroencephalographic Density Spectrum Array During Deep Sedation in High Risk Patients.
Brief Title: EEG Spectral Pattern of Deep Sedation-induced Airway Adverse Effects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202209055DINB
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Procedural Sedation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Geriatric population: patient with ages above 65-yr
  Interventions: Diagnostic Test: Airmod breathing sound monitoring
- Pediatric population: patient with ages between 4-8 year old
  Interventions: Diagnostic Test: Airmod breathing sound monitoring

INTERVENTIONS:
Diagnostic Test: Airmod breathing sound monitoring — Respiratory monitoring and sedation depth monitoring will be applied during procedural sedation.
  Other Names: Electroencephalographic monitoring; Capnographic monitoring

SUMMARY:
To investigate the associations bewteen the sedation level and the airway adverse effects by using the EEG, Airmod breath sound monitor and the capnography.

DETAILED DESCRIPTION:
Deep sedation is mandatory for many invasive procedures such as the digestive endoscopy, bronchoscopy and cystoscopy. However, deep sedation may induce respiratory adverse effects including airway obstruction, hypoventilation and apnea. These respiratory adverse effects, which may occur in more than 20% of high-risk groups (eg, children, the elderly, and patients with sleep apnea), hence, are the major concerns of the anesthetic care. However, It is difficult for clinicians to objectively quantify the sedation level and find the associations of inadequate sedation level and the occurrence of respiratory adverse effects.

Airway obstruction and respiratory rate decline during deep sedation are conventionally monitored by using capnography(EtCO2 waveform). However, previous studies have tracheal breath sound monitoring can achieve better detection accuracy than the capnography. The novel Airmod smart breathing monitor has the functions of breath sound recording, anti-noise signal processing, event recording and respiratory rate analysis and research. Through the continuous breath sound recording, airway adverse effects during sedation may be detected, and these breathing spectrogram can be presented for image analysis. This is helpful for researcher to identify associations between airway adverse effect and the sedation level.

The state-of-art anesthetic depth is determined by using the electroencephalogram (EEG). Both EEG raw data or the EEG spectrogram graphs may be used for quantify the sedation level with respiratory adverse effects. Accordingly, this study aims to investigate the associations between the sedation level and the airway adverse effects by using the EEG monitor, Airmod breath sound monitor and the capnography.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing procedural sedation with expected produre time longer than 30 minutes

* Pediatric group: age 4-8 year-old
* Geriatric group: age>= 65 year-old

Exclusion Criteria:

* Preoperative active brain conditions (dementia, Parkinsonism, seizure)
* A history of nasal or oral tumor

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two patient groups of higher risk for invasive procedural sedation will be investigated, namely the pediatric patients and geriatric patients.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Occurence of airway obstruction during sedation | 0.5-2 hours
  Airway obstruction detected by the breath sound monitor or capnography
Occurence of apnea event during sedation | 0.5-2 hours
  Apnea detected by the breath sound monitor or capnography

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The IPD can be obtained by contacting the corresponding author after the study is published
Supporting Information: CSR
Time Frame: The data will be availabel after publication.
Access Criteria: For research purpose only. The IPD will not be provided for commercial purpose.